CLINICAL TRIAL: NCT00486642
Title: A Phase 2 Study of GW786034 (Pazopanib) With or Without Bicalutamide in Hormone Refractory Prostate Cancer
Brief Title: Pazopanib Hydrochloride With or Without Bicalutamide in Treating Patients With Prostate Cancer That Did Not Respond to Hormone Therapy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00200; NCI-2009-00200 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); PMH-PHL-058; PMH-10036920; CDR0000549528; PHL-058 (Other: University Health Network-Princess Margaret Hospital); 7640 (Other: CTEP); N01CM00032 (NIH); N01CM62203 (NIH)
Record Dates: First submitted 2007-06-13; First posted 2007-06-14 (Estimated); Results first posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-04

CONDITIONS: Hormone-Resistant Prostate Cancer; Recurrent Prostate Carcinoma
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bicalutamide; pazopanib

ARMS (2):
- Arm A (pazopanib hydrochloride) (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-28.
  .
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pazopanib Hydrochloride; Other: Pharmacological Study
- Arm B (pazopanib hydrochloride, bicalutamide) (Experimental): Patients receive pazopanib hydrochloride PO QD on days 1-28. Patients also receive bicalutamide PO QD on days 8-28 of course 1 and on days 1-28 in all subsequent courses.
  Interventions: Drug: Bicalutamide; Other: Laboratory Biomarker Analysis; Drug: Pazopanib Hydrochloride; Other: Pharmacological Study

INTERVENTIONS:
Drug: Bicalutamide — Given PO
  Other Names: Casodex; Cosudex; ICI 176,334; ICI 176334
  Arms: Arm B (pazopanib hydrochloride, bicalutamide)
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pazopanib Hydrochloride — Given PO
  Other Names: GW786034B; Votrient
Other: Pharmacological Study — Correlative studies

SUMMARY:
This randomized phase II trial is studying how well giving pazopanib with or without bicalutamide works in treating patients with prostate cancer that did not respond to hormone therapy. Pazopanib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the tumor. Androgens can cause the growth of prostate cancer cells. Antihormone therapy, such as bicalutamide, may lessen the amount of androgens made by the body. Giving pazopanib hydrochloride together with bicalutamide may be an effective treatment for prostate cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the therapeutic activity of GW786034 (pazopanib hydrochloride) with and without bicalutamide in the treatment of hormone-refractory prostate cancer using prostate specific antigen (PSA)-response rate.

SECONDARY OBJECTIVES:

I. To estimate objective tumor response in patients with measurable disease. II. To estimate the median time to progression. III. To investigate the safety and tolerability of GW786034 with and without bicalutamide.

IV. To estimate the median duration of PSA-response. V. To determine the steady state levels of GW786034 with and without bicalutamide.

VI. To investigate the correlation between prior exposure to bicalutamide and non-steroidal anti-androgens with response and survival outcomes.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive pazopanib hydrochloride orally (PO) once daily (QD) on days 1-28.

ARM II: Patients receive pazopanib hydrochloride PO QD on days 1-28. Patients also receive bicalutamide PO QD on days 8-28 of course 1 and on days 1-28 in all subsequent courses.

Courses in both arms repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 4 weeks for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed prostate cancer
* Must have received prior hormonal therapy, including either medical (luteinizing hormone-releasing hormone [LHRH] agonist) or surgical (orchiectomy) castration

  * Castrate level of testosterone (< 50 ng/dL)
  * Patients treated with LHRH agonists must continue or restart this therapy
* Must have radiological documentation of either measurable or non-measurable disease
* Must show documented progression of prostate cancer while on hormonal therapy as indicated by PSA increase

  * Rising PSA is defined as ≤ 2 consecutive rises in PSA taken ≥ 1 week and ≤ 2 months apart
* PSA >= 5 ng/mL
* No known brain metastases
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Life expectancy > 3 months
* White blood cell (WBC) >= 3,000/mm^3
* Absolute neutrophil count (ANC) >= 1,500/mm^3
* Platelet count >= 100,000/mm^3
* International normalized ratio (INR) =< 1.2
* Activated partial thromboplastin time (PTT) =< 1.2 times upper limit of normal (ULN)
* Bilirubin normal
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) =< 1.5 times ULN
* Creatinine normal OR creatinine clearance >= 60 mL/min
* Fertile patients must use effective contraception
* No history of allergic reactions attributed to compounds of similar chemical or biological composition to pazopanib hydrochloride or bicalutamide
* Proteinuria =< 1+ on 2 consecutive dipsticks taken >= 1 week apart
* QTc < 480 msec
* No significant electrocardiogram (ECG) abnormalities
* No poorly controlled hypertension (systolic blood pressure [BP] > 150 mm Hg or diastolic BP > 90 mm Hg)
* No condition (e.g., gastrointestinal [GI] tract disease resulting in an inability to take oral medication or a requirement for intravenous (IV) alimentation; prior surgical procedures affecting absorption; or active peptic ulcer disease) that impairs the ability to swallow and retain pazopanib hydrochloride tablets
* No serious or nonhealing wound, ulcer, or bone fracture
* No abdominal fistula, gastrointestinal (GI) perforation, or intra-abdominal abscess within the past 28 days
* No cerebrovascular accident within the past 6 months
* No myocardial infarction, cardiac arrhythmia, admission for unstable angina, cardiac angioplasty, or stenting within the past 12 weeks
* No venous thrombosis within the past 12 weeks
* No New York Heart Association (NYHA) class III-IV heart failure

  * Patients with a history of NYHA class II heart failure who are asymptomatic on treatment are eligible
* No concurrent uncontrolled illness, including, but not limited to, ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* Recovered from all prior therapy
* Prior neoadjuvant or adjuvant chemotherapy allowed
* More than 4 weeks since prior chemotherapy (6 weeks for nitrosoureas or mitomycin C) or radiotherapy
* At least 4 weeks since prior antiandrogens
* At least 4 weeks since prior surgery
* No prior bicalutamide therapy lasting > 3 months in duration
* Concurrent steroids allowed if no change in steroid dosage within the past 4 weeks
* No other concurrent investigational agents
* No concurrent therapeutic warfarin

  * Concurrent low molecular weight heparin or prophylactic low-dose warfarin allowed
* No concurrent combination antiretroviral therapy for human immunodeficiency virus (HIV)-positive patients

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2007-09; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kim Chi, Principal Investigator — University Health Network-Princess Margaret Hospital
Locations (6):
- Canada (6):
  - BCCA-Vancouver Cancer Centre, Vancouver, British Columbia
  - Juravinski Cancer Centre at Hamilton Health Sciences, Hamilton, Ontario
  - Cancer Centre of Southeastern Ontario at Kingston General Hospital, Kingston, Ontario
  - London Regional Cancer Program, London, Ontario
  - Ottawa Hospital and Cancer Center-General Campus, Ottawa, Ontario
  - University Health Network-Princess Margaret Hospital, Toronto, Ontario

REFERENCES:
- [Derived] Sridhar SS, Joshua AM, Gregg R, Booth CM, Murray N, Golubovic J, Wang L, Harris P, Chi KN. A phase II study of GW786034 (pazopanib) with or without bicalutamide in patients with castration-resistant prostate cancer. Clin Genitourin Cancer. 2015 Apr;13(2):124-9. doi: 10.1016/j.clgc.2014.06.001. Epub 2014 Jun 8. PMID 24993934

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (Pazopanib): Arm I - Patients receive pazopanib hydrochloride PO QD on days 1-28.
  Laboratory Biomarker Analysis: Correlative studies
  Pazopanib Hydrochloride: Given PO
  Pharmacological Study: Correlative studies
- Arm II (Pazopanib & Bicalutamide): Arm II - Patients receive pazopanib hydrochloride PO QD on days 1-28. Patients also receive bicalutamide PO QD on days 8-28 of course 1 and on days 1-28 in all subsequent courses.
Period: Overall Study
Arm/Group | Arm I (Pazopanib) | Arm II (Pazopanib & Bicalutamide)
Started | 10 | 13
Completed | 10 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Arm A - Pazopanib: Patients receive pazopanib hydrochloride PO QD on days 1-28.
  Laboratory Biomarker Analysis: Correlative studies
  Pazopanib Hydrochloride: Given PO
  Pharmacological Study: Correlative studies
- Arm B - Pazopanib + Bicalutamide: Patients receive pazopanib hydrochloride PO QD on days 1-28. Patients also receive bicalutamide PO QD on days 8-28 of course 1 and on days 1-28 in all subsequent courses.
  Laboratory Biomarker Analysis: Correlative studies
  Pazopanib Hydrochloride: Given PO
  Pharmacological Study: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Arm A - Pazopanib | Arm B - Pazopanib + Bicalutamide | Total
Number analyzed (Participants) | 10 | 13 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 12
  >=65 years | 2 | 9 | 11
Age, Continuous [Median (Full Range); unit: years] | 71 [54 to 77] | 70 [51 to 85] | 71 [51 to 85]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 10 | 13 | 23
Region of Enrollment [Number; unit: participants]
  Canada | 10 | 13 | 23

OUTCOME MEASURES:

1. Primary Outcome: PSA Response Rate
Description: Prostate-specific antigen (PSA) response rate (defined as a confirmed > / = 50% decline (minimum 5ng/ml) in PSA from baseline maintained for >4 weeks, and without other evidence of disease progression documented at time of confirmatory values).
Time Frame: Up to 12 weeks
Population: 9 evaluable in Arm A + 12 evaluable in Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Pazopanib | Arm B - Pazopanib + Bicalutamide
Number analyzed (Participants) | 9 | 12
Participants | 1 | 2

2. Secondary Outcome: Objective Tumor Response Rate as Assessed by RECIST Criteria
Description: RECIST PR defined as - At least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Time from start of treatment to time criteria are met for disease progression or death from any cause, whichever came first, assessed up to 5 years
Population: 5 evaluable patients in Arm A + 9 evaluable patients in Arm B
Measure: Number; unit: patient
Arm/Group | Arm A - Pazopanib | Arm B - Pazopanib + Bicalutamide
Number analyzed (Participants) | 5 | 9
patient | 0 | 1

3. Secondary Outcome: Progression-free Survival
Description: PFS is defined as the time from treatment initiation to disease progression or death from any cause, whichever came first.
  Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions
Time Frame: From time of treatment initiation to disease progression or death from any cause, whichever came first, assessed up to 5 years
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Pazopanib | Arm B - Pazopanib + Bicalutamide
Number analyzed (Participants) | 10 | 13
months | 7.3 [1.2 to NA] — Not reached | 11.3 [4.84 to NA] — Not reached

4. Secondary Outcome: Median Duration of PSA-Response
Description: Definition of PSA response: >= 50% fall (minimum 5 ng/ml) in PSA from baseline maintained for >4 weeks, and without other evidence of disease progression documented at time of confirmatory values.
  PSA response duration will commence on the date of the first >=50% decline in PSA. The response duration ends when PSA progression criteria are met with the second increasing PSA value.
  PSA progression in PSA responders: rise in PSA of 50% (minimum 5ng/ml) above nadir value and confirmed by a second increasing value at least 1 week later.
Time Frame: From time PSA response criteria are met until time PSA progression criteria are met or death from any cause, whichever came first, up to 5 years
Population: 1 patient in Arm A and 2 patients in Arm B had a PSA response.
Measure: Median (Full Range); unit: months
Arm/Group | Arm A - Pazopanib | Arm B - Pazopanib + Bicalutamide
Number analyzed (Participants) | 1 | 2
months | 8.3 [8.3 to 8.3] | 13.1 [2.3 to 23.9]

5. Secondary Outcome: Stable Disease Rate as Assessed by RECIST Criteria
Description: RECIST Stable defined as - Neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum diameters while on study.
Time Frame: Measured from the start of the treatment until the criteria for progression are met or death from any cause, whichever came first, assessed up to 5 years
Population: 5 evaluable patients in Arm A + 9 evaluable patients in Arm B
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A - Pazopanib | Arm B - Pazopanib + Bicalutamide
Number analyzed (Participants) | 5 | 9
Participants | 2 | 8

6. Secondary Outcome: Time to Disease Progression
Description: Earliest date on which disease progression was determined by any of the methods listed: PSA progression, objective disease progression (Response Evaluation Criteria in Solid Tumors [RECIST] criteria) or cancer-related symptomatic progression.
Time Frame: as for outcome 2
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A - Pazopanib | Arm B - Pazopanib + Bicalutamide
Number analyzed (Participants) | 10 | 13
months | 7.3 [1.20 to NA] — Not reached | 11.3 [4.84 to NA] — Not reached

7. Secondary Outcome: Toxicity
Description: Patients who came off treatment due to toxicity.
Time Frame: Assessed up to 5 years
Measure: Number; unit: participants
Groups:
- Arm A (Pazopanib): Patients receive pazopanib hydrochloride PO QD on days 1-28.
  Laboratory Biomarker Analysis: Correlative studies
  Pazopanib Hydrochloride: Given PO
  Pharmacological Study: Correlative studies
- Arm B (Pazopanib + Bicalutamide): Patients receive pazopanib hydrochloride PO QD on days 1-28. Patients also receive bicalutamide PO QD on days 8-28 of course 1 and on days 1-28 in all subsequent courses.
  Laboratory Biomarker Analysis: Correlative studies
  Pazopanib Hydrochloride: Given PO
  Pharmacological Study: Correlative studies
Arm/Group | Arm A (Pazopanib) | Arm B (Pazopanib + Bicalutamide)
Number analyzed (Participants) | 10 | 13
participants | 3 | 6

8. Other Pre Specified Outcome: Median Survival Time
Description: Calculated by Kaplan and Meier
Time Frame: Up to 1 year after completion of treatment
Population: Very little death information is captured for this study so OS analysis was not done.
Arm/Group | Arm A - Pazopanib | Arm B - Pazopanib + Bicalutamide
Number analyzed (Participants) | 0 | 0

9. Other Pre Specified Outcome: Survival Rate
Description: Calculated by Kaplan and Meier.
Time Frame: At 1 year
Population: Very little death information is captured for this study so OS analysis was not done.
Arm/Group | Arm A - Pazopanib | Arm B - Pazopanib + Bicalutamide
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Arm A - Pazopanib | Arm B - Pazopanib + Bicalutamide
All-Cause Mortality (participants affected / at risk) | 1/10 | 2/13
Serious Adverse Events (participants affected / at risk) | 2/10 | 3/13
Other Adverse Events (participants affected / at risk) | 10/10 | 13/13
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A - Pazopanib (N=10) | Arm B - Pazopanib + Bicalutamide (N=13)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 1 (1) | 1 (1)
Fever (General disorders) | 1 (1) | 0 (0)
Hematuria (Renal and urinary disorders) | 1 (2) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Erectile dysfunction (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Glucose intolerance (Metabolism and nutrition disorders) | 0 (0) | 1 (2)
Urinary frequency (Renal and urinary disorders) | 0 (0) | 1 (1)
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (1)
Lymphocyte count decreased (Investigations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A - Pazopanib (N=10) | Arm B - Pazopanib + Bicalutamide (N=13)
Abdominal distension (Gastrointestinal disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Acidosis (Metabolism and nutrition disorders) | 0 | 2
Acoustic nerve disorder NOS (Nervous system disorders) | 0 | 1
Activated partial thromboplastin time prolonged (Investigations) | 0 | 1
Agitation (Psychiatric disorders) | 0 | 1
Alanine aminotransferase increased (Investigations) | 6 | 5
Alkaline phosphatase increased (Investigations) | 7 | 5
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Anal mucositis (Gastrointestinal disorders) | 0 | 1
Anemia (Blood and lymphatic system disorders) | 7 | 12
Anorexia (Metabolism and nutrition disorders) | 7 | 9
Anxiety (Psychiatric disorders) | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 5 | 4
Aspartate aminotransferase increased (Investigations) | 5 | 7
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 4 | 5
Bladder infection (Infections and infestations) | 1 | 0
Blood and lymphatic system disorders - Other (Blood and lymphatic system disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 4 | 4
Blurred vision (Eye disorders) | 0 | 1
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 2
Chest pain - cardiac (Cardiac disorders) | 0 | 1
Chills (General disorders) | 2 | 1
Confusion (Psychiatric disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 2 | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Creatinine increased (Investigations) | 1 | 5
Dehydration (Metabolism and nutrition disorders) | 0 | 1
Depression (Psychiatric disorders) | 1 | 1
Diarrhea (Gastrointestinal disorders) | 5 | 9
Dizziness (Nervous system disorders) | 0 | 7
Dry mouth (Gastrointestinal disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 2 | 1
Dyspepsia (Gastrointestinal disorders) | 4 | 3
Dysphasia (Nervous system disorders) | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 | 4
Edema limbs (General disorders) | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 1
Fatigue (General disorders) | 9 | 11
Fever (General disorders) | 1 | 1
Flatulence (Gastrointestinal disorders) | 2 | 0
Flu like symptoms (General disorders) | 0 | 1
Flushing (Vascular disorders) | 2 | 1
Fracture (Injury, poisoning and procedural complications) | 0 | 1
Gait disturbance (General disorders) | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 1
Gastrointestinal disorders - Other (Gastrointestinal disorders) | 1 | 2
General disorders and administration site conditions - Other (General disorders) | 0 | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
GGT increased (Investigations) | 0 | 1
Gingival pain (Gastrointestinal disorders) | 0 | 1
Glucose intolerance (Metabolism and nutrition disorders) | 0 | 1
Headache (Nervous system disorders) | 1 | 3
Hematoma (Vascular disorders) | 1 | 1
Hematuria (Renal and urinary disorders) | 3 | 2
Hemoglobinuria (Renal and urinary disorders) | 4 | 3
Hemorrhoids (Gastrointestinal disorders) | 1 | 1
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hot flashes (Vascular disorders) | 4 | 4
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 2
Hypermagnesemia (Metabolism and nutrition disorders) | 0 | 1
Hypertension (Vascular disorders) | 8 | 10
Hypoalbuminemia (Metabolism and nutrition disorders) | 5 | 6
Hypocalcemia (Metabolism and nutrition disorders) | 2 | 1
Hypoglycemia (Metabolism and nutrition disorders) | 1 | 1
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 3 | 4
Hyponatremia (Metabolism and nutrition disorders) | 3 | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 2
Hypotension (Vascular disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 1
Insomnia (Psychiatric disorders) | 1 | 2
Ischemia cerebrovascular (Nervous system disorders) | 0 | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 0 | 1
Lymphocyte count decreased (Investigations) | 7 | 9
Memory impairment (Nervous system disorders) | 0 | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 0 | 1
Mucositis oral (Gastrointestinal disorders) | 2 | 3
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 1
Musculoskeletal and connective tissue disorder - Other (Musculoskeletal and connective tissue disorders) | 2 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 2
Nausea (Gastrointestinal disorders) | 1 | 7
Nervous system disorders - Other (Nervous system disorders) | 0 | 1
Neutrophil count decreased (Investigations) | 4 | 4
Non-cardiac chest pain (General disorders) | 1 | 0
Oral pain (Gastrointestinal disorders) | 0 | 1
Pain (General disorders) | 3 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 | 4
Pelvic pain (Reproductive system and breast disorders) | 0 | 1
Penile infection (Infections and infestations) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 1
Platelet count decreased (Investigations) | 4 | 6
Proteinuria (Renal and urinary disorders) | 4 | 9
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Pulmonary fibrosis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 4
Rectal hemorrhage (Gastrointestinal disorders) | 2 | 2
Rectal pain (Gastrointestinal disorders) | 0 | 1
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 3
Respiratory, thoracic and mediastinal disorders - Other (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Sinus bradycardia (Cardiac disorders) | 0 | 1
Sinus pain (Nervous system disorders) | 0 | 1
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 1 | 1
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 | 0
Stomach pain (Gastrointestinal disorders) | 0 | 1
Tinnitus (Ear and labyrinth disorders) | 0 | 1
Tooth infection (Infections and infestations) | 0 | 3
Toothache (Gastrointestinal disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Upper respiratory infection (Infections and infestations) | 3 | 1
Urinary frequency (Renal and urinary disorders) | 2 | 6
Urinary incontinence (Renal and urinary disorders) | 0 | 2
Urinary retention (Renal and urinary disorders) | 1 | 1
Urinary tract pain (Renal and urinary disorders) | 0 | 1
Vascular disorders - Other (Vascular disorders) | 0 | 1
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Vomiting (Gastrointestinal disorders) | 1 | 6
Watering eyes (Eye disorders) | 1 | 0
Weight loss (Investigations) | 1 | 6
White blood cell decreased (Investigations) | 4 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less